CLINICAL TRIAL: NCT03054961
Title: Cerebral Oxygen Saturation and Cytochrome Oxidase REDOX State in Children With Epilepsy: A Pilot Study - Multichannel Near-infrared Spectroscopy (NIRS) for Epilepsy Seizure Detection
Brief Title: Cerebral Oxygen Saturation and Cytochrome Oxidase REDOX State in Children With Epilepsy: A Pilot Study
Status: Completed | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Marquette University (Other)
Responsible Party: Principal Investigator, Rene Andrade-Machado, Assistant Professor, Medical College of Wisconsin
Other Study IDs: PRO00046065
Record Dates: First submitted 2017-02-10; First posted 2017-02-16 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Epilepsies, Partial
Keywords: epilepsy; cytochrome oxidase redox state; childhood epilepsy; partial epilepsy; NIRS; near-infrared spectroscopy; regional cerebral oxygen saturation
MeSH Terms: conditions — Epilepsies, Partial; Epilepsy | interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Epilepsy patients: Near-infrared spectroscopy for subjects with partial (focal) epilepsy seizures being studied in the EMU.
  Interventions: Device: Near-infrared spectroscopy

INTERVENTIONS:
Device: Near-infrared spectroscopy — Measurement of CCO redox state and cerebral oxygenation during epileptic seizures.

SUMMARY:
The purpose of this pilot study is to describe the relationship of regional cerebral oximetry and cytoximetry, measured using near-infrared spectroscopy, with seizure activity in the periictal period in children with epilepsy.

DETAILED DESCRIPTION:
Pediatric subjects with partial (focal) epilepsy seizure disorders will be studied using near-infrared spectroscopy for cytochrome c oxidase (CCO) redox state and blood oxygen saturation. Along with routine EEG monitoring, a set of light sensors, called optodes, attached to a net/cap/device that goes over the head will be put on. These optodes will send out very weak red light signals, which will pass through the scalp and bounce back to detectors on the netting. The changes in the light signals will be used to calculate the changes in the various forms of the enzyme CCO, as well as the amount of oxygen in the blood. We hope to use these measurements to study changes in blood flow and cellular energy usage in the brain during seizures, which might help us to understand epilepsy better in the future and design better treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric epilepsy patients who can provide assent (lower limit age 7).
2. Diagnosis of partial (focal) epilepsy and/or frequent interictal spike activity on EEG.
3. Clinical EEG supporting diagnosis of partial(focal) epilepsy and/or frequent interictal spike activity

Exclusion Criteria:

1. History of unrepaired or palliated congenital cyanotic heart disease
2. History of traumatic head injury or head wounds to the extent that precludes safe and consistent placement of NIRS-EEG probes.
3. Guardian does not give consent or patient is unable to consent/assent to participate in the study
4. Clinical care provider or investigator determines the patient is not appropriate candidate for the study
5. Lack of current seizure care plan in Children's Hospital medical record
6. Known sensitivity or allergy to EEG gel

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study subjects will include pediatric patients from 7 and older with a known seizure disorder. This study design is a prospective observational case-control where the subjects are their own controls. This is accomplished by comparing brain regions of electrical spikes to regions without spikes as measured by EEG and NIRS during resting state, structured task paradigm completion and, if seizure activity incidentally occurs during the study visit, NIRS data from brain regions of electrical spikes from seizure activity will be compared to other brain regions.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2017-02-10 (Actual); Primary Completion 2023-06-07 (Actual); Study Completion 2023-06-07 (Actual)

PRIMARY OUTCOMES:
Change in CCO redox state and oxygen saturation | 1 week
  Regional cerebral saturation of oxygen and/or cytochrome oxidase redox state will change prior, during, and after onset of seizure activity when compared to non-seizure side of brain.

CONTACTS AND LOCATIONS:
Overall Officials: Rene Andrade-Machado, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- The Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No